CLINICAL TRIAL: NCT03504579
Title: Real-time fMRI Feedback as a Tool to Mitigate Auditory Hallucinations in Schizophrenia
Brief Title: Rt-fMRI Neurofeedback and AH in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Margaret Niznikiewicz, associate professor; lab director, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 7304878-01
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Audio Visual Hallucinations; Neurofeedback; Schizophrenia; Superior Temporal Gyrus
Keywords: rt-fMRI; MRI; schizophrenia; auditory hallucinations; neurofeedback
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Intervention Model Description: In the R61 phase of the study,changes in a target brain region(s) will be demonstrated after the rt-fMRI based neurofeedback session.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rt-fMRI neurofeedback aimed at STG (Experimental): One session of rt-fMRI neurofeedback from the patient's STG.
  Interventions: Other: rt-fMRI neurofeedback
- sham rt-fMRI (Sham Comparator): One session of rt-fMRI neurofeedback from the patient's motor cortex.
  Interventions: Other: rt-fMRI neurofeedback

INTERVENTIONS:
Other: rt-fMRI neurofeedback — use of real time fMRI neurofeedback to achieve targeted brain changes

SUMMARY:
Auditory hallucinations in schizophrenia are one of the major symptoms of this disease and a major source of psychological discomfort. They are often difficult or impossible to treat with existing methods. This study will test the use of real-time fMRI neurofeedback to mitigate auditory verbal hallucinations in patients whose hallucinations are resistant to medication. Half of the patients will receive real time fMRI neurofeedback from a brain region involved in auditory hallucinations and half will receive it from motor cortex.

DETAILED DESCRIPTION:
Auditory verbal hallucinations (AH) have long been a hallmark of schizophrenia (SZ) and are one of its major diagnostic features. They are difficult to manage with existing treatment options. Here, neurofeedback will be used to regulate the superior temporal gyrus (STG) activation which will not only lead to activation changes in the STG, but also to changes in the default mode network (DMN).

The investigators will study SZ patients with medication resistant AH in the rt-fMRI intervention arm and in the sham-rt-fMRI arm. In both arms, the task and the rt-fMRI session structure will be identical. The SZ-intervention group will receive feedback from the STG while SZ-sham group will receive feedback from the motor cortex. In addition, 2 functional fMRI tasks will examine the effect of rt-fMRI neurofeedback and of sham-rt-fMRI on brain response.

The investigators will randomly assign 48 SZ patients to either SZ-intervention (n=24) or SZ-sham-rtfMRI (n=24). The STG targeted neurofeedback is predicted to bring changes in brain regions involved in AH (STG and DMN) in SZ-intervention group only. The R61 GO criterion will be BOLD signal reduction in the STG, and resting state connectivity reduction between MPFC-PCC, post rt-fMRI-feedback in SZ-intervention group.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of schizophrenia or schizoaffective disorder based on SCID interview (DSM-5) and
* the presence of auditory hallucinations (PANSS, item 3, score ≥4) with frequency of AH being at least once daily;
* age between 18-55 years;
* estimated IQ of above 80 as measured by WASI;
* English as the primary language;
* right-handed as determined by the Edinburgh Handedness Inventory (scoring + 60; Oldfield, 1971);
* an ability and desire to participate in the testing program as explained by an experimenter and confirmed with a written consent form.

Exclusion Criteria:

* history of ECT for the last 5 years;
* history of neurological illness or a traumatic head injury, defined as loss of consciousness for more than 5 minutes and/or structural sequelae following head trauma;
* history of severe or moderate alcohol (AUD) or substance use disorder (SUD) in the past five years, or mild AUD or SUD within the last year, according to DSM-5;
* the use, in the preceding year of steroids or barbiturates, which can affect cognitive function;
* hearing, vision or upper body impairment
* alcohol use in the last 24 hours;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
rt-fMRI neurofeedback from STG | 1-2 weeks, post rt-fMRI session
  changes in BOLD activation in STG

SECONDARY OUTCOMES:
rt-fMRI neurofeedback from mPFC | 1-2 weeks, post rt-fMRI session
  changes in BOLD activation in mPFC

CONTACTS AND LOCATIONS:
Overall Officials: margaret niznikiewicz, ph.d, Principal Investigator — VA Boston Healthcare System; susan whitfield-Gabrieli, Ph.D., Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Veterans Administration Health Care System, Brockton, Massachusetts, United States

REFERENCES:
- [Derived] Zhang J, Tusuzian E, Morfini F, Bauer CCC, Stone L, Awad A, Shinn AK, Niznikiewicz MA, Whitfield-Gabrieli S. Brain Structural and Functional Neuroimaging Features are Associated With Improved Auditory Hallucinations in Patients With Schizophrenia After Real-Time fMRI Neurofeedback. Depress Anxiety. 2025 Apr 8;2025:2848929. doi: 10.1155/da/2848929. eCollection 2025. PMID 40236821
- [Derived] Morfini F, Bauer CCC, Zhang J, Whitfield-Gabrieli S, Shinn AK, Niznikiewicz MA. Targeting the superior temporal gyrus with real-time fMRI neurofeedback: A pilot study of the indirect effects on self-referential processes in schizophrenia. Schizophr Res. 2024 Aug;270:358-365. doi: 10.1016/j.schres.2024.06.036. Epub 2024 Jul 4. PMID 38968807